CLINICAL TRIAL: NCT05760014
Title: Interest of Medical Hypnosis in Reducing Stress and Improving the Experience of Hospitalization in Internal Medicine
Brief Title: Medical Hypnosis and Stress Reduction in Hospitalization
Acronym: HYPNOSTRESS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_0670; 2022-A02406-37 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2023-02-24; First posted 2023-03-08 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Stress
Keywords: hypnosis; perceived stress; place of safety; case control study

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAS patients: CAS patients with a conventional follow-up who will benefit from the hypnosis technique known as "Place of Safety" on their admission to conventional hospitalization.
- TEMOINS patients: TEMOINS patients with conventional follow-up who will not benefit from the medical hypnosis technique.

SUMMARY:
Patients with chronic diseases, especially rare diseases with uncertain diagnoses, have a representation of their disease and an experience of their hospitalization that is sometimes traumatic, distressing and painful. Patients hospitalized can benefit from non-medicinal techniques, such as medical hypnosis, which could improve the perceived stress in these patients and thus optimize the hospitalization experience. The aim of this study is to evaluate the impact of medical hypnosis in reducing stress and improving the experience of hospitalization comparing two groups : a group (cases) benefiting from an hypnotic technic " the place of safety " and a control group without intervention during hospitalization

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalised in the internal medicine department of the Lille University Hospital
* Age>= 18 years
* Patients having expressed their non opposition

Exclusion Criteria:

* Not covered by the social security system
* Person unable to receive informed information
* Persons deprived of liberty
* Persons under legal protection (guardianship / curatorship)
* Psychotic and/or dementia disorders
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised for their chronic illness
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
STAI questionnaire dimension STAI completed at discharge. | At discharge, an average 10 days
  STAI-ETAT

SECONDARY OUTCOMES:
The STAI ETAT (the current emotional state) questionnaire | at baseline and at discharge, an average 10 days
  State Trait Anxiety Inventory Etat - Trait (40 questions - each item has a score from 1 to 4 (4 being the highest level of anxiety))
The STAI-TRAIT (the usual emotional state ) questionnaire | at baseline and at discharge, an average 10 days
  State-Trait Anxiety Inventory (STAI-TRAIT) SCORE: 20 items in the form of a 4-response Likert scale (from 1 : low anxiety to 4 : highest anxiety). The score goes from 20 to 80 depending of the degree of anxiety
patient opinion questionnaire | At discharge, an average 10 days
The difference in STAI STATUS score between the questionnaire completed post-hypnotic treatment and the questionnaire at admission | At discharge, an average 10 days
The ordinal severity scale correlated with the STAI ETAT questionnaire score; | At discharge, an average 10 days
Self-rated stress scale correlated with the STAI ETAT questionnaire score. | At discharge, an average 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Mereym-Maud FAHRAT, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- service de médecine interne CHU Lille, Lille, France